CLINICAL TRIAL: NCT05321914
Title: The Impact of the Time of Day on Metabolic Responses to Resistance Exercise in Adults Who Are Obese or Overweight: a Randomised Controlled Trial
Brief Title: Resistance Exercise, Metabolism and Time of Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200210068
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Disease
Keywords: exercise; muscle; metabolism; circadian
MeSH Terms: conditions — Metabolic Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Habitual physical activity
- Morning exercise (Experimental): Exercise training in the morning (6:00-10:00am)
  Interventions: Behavioral: Exercise training
- Evening exercise (Experimental): Exercise training in the evening (4:00-8:00pm)
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Exercise will consist of 1 set x 9 exercises x 3 sessions per week x 6 weeks. The load to be used during training will be calculated as 80% of one-repetition maximum (1RM) with each set performed to failure. 1RM will be re-tested on week 3, and the load adjusted accordingly, and upon completion of the study. During the training period, all sessions of training will be supervised by the researcher. The following exercises will be performed: Bench press, biceps curl, lat pull down, overhead press, lateral raise, leg extension, leg curl and calf raise.
  Arms: Evening exercise; Morning exercise

SUMMARY:
The aim of the current study is to determine the effect of time of day on the muscle and metabolic responses to resistance exercises in obese or overweight adults. To achieve this aim we have the following objectives:

1. Compare the effects of resistance exercise training performed in the morning vs the evening on insulin sensitivity
2. Compare the effects of resistance exercise training performed in the morning vs the evening on gains in muscle mass and strength
3. Compare the acute glucose responses to resistance exercise performed in the morning vs the evening

ELIGIBILITY:
Inclusion Criteria:

* pass the physical activity readiness questionnaire
* body mass index (BMI) >27kg/m² and limited to 40 kg/m².

Exclusion Criteria:

* Prior surgery for weight loss
* Prior history of heart, lung, cancer, endocrine or liver disease
* Participating in more than 1 hour structured exercise training per week

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Change from baseline to 6 weeks
  Insulin sensitivity calculated via the Matsuda Index during an oral glucose tolerance test

SECONDARY OUTCOMES:
Change in vastus lateralis muscle thickness | Change from baseline to 6 weeks
  Muscle thickness of the vastus lateralis muscle measured via ultrasound
Change in whole body lean mass | Change from baseline to 6 weeks
  whole body lean mass measured via bio-electrical impedance
Change in whole body fat mass | Change from baseline to 6 weeks
  whole body fat mass measured via bio-electrical impedance
Change in one-repetition maximum muscle strength | Change from baseline to 6 weeks
  Sum of one-repetition maximum of Bench press, biceps curl, lat pull down, overhead press, lateral raise, leg extension, leg curl and calf raise exercise
Change in knee extensor maximal isometric torque | Change from baseline to 6 weeks
  Knee extensor maximal isometric torque measured during a maximal voluntary contraction
Change in grip strength | Change from baseline to 6 weeks
  Grip strength measured with a hand held dynamometer
Change in mean glucose levels | Change from baseline to 6 weeks
  Mean glucose levels measured via continuous glucose monitors
Change in glucose variability | Change from baseline to 6 weeks
  Glucose variability measured via continuous glucose monitors

CONTACTS AND LOCATIONS:
Locations (1):
- Stuart Robert Gray, Glasgow, United Kingdom

REFERENCES:
- [Derived] Dighriri A, Lithgow H, Gabriel B, Altuwrqi M, Dunning E, Johnston L, Boyle JG, Logan G, Gray SR. The impact of the time of day on muscle and metabolic responses to resistance exercise in healthy adults: A randomised controlled trial. Exp Physiol. 2025 Nov 13. doi: 10.1113/EP093020. Online ahead of print. PMID 41231202